CLINICAL TRIAL: NCT05330702
Title: Ultrasound-based Imaging to Detect Early Changes of Hard and Soft Tissue Around Immediately Placed Implants With or Without Soft Tissue Augmentation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforeseen Event - Original PI left the University of Iowa
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Shaoping Zhang, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202203162
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-08

CONDITIONS: Tooth Extraction; Immediate Implant Placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Tuberosity Connective Tissue Graft (CTG) (Experimental): Subjects in this arm will have a tuberosity connective tissue graft at the time of immediate implant placement.
  Interventions: Procedure: Tuberosity Connective Tissue Graft (CTG)
- Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft (Experimental): Subjects in this arm will have Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft at the time of immediate implant placement.
  Interventions: Device: Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft No Intervention: No Soft Tissue Augmentation
- No Soft Tissue Augmentation (No Intervention): Subjects in this arm will have no soft tissue augmentation at the time of immediate implant placement.

INTERVENTIONS:
Device: Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft No Intervention: No Soft Tissue Augmentation — Fibro-gide is the VCMX
  Other Names: Fibro-Gide, Geistlich Pharma
  Arms: Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft
Procedure: Tuberosity Connective Tissue Graft (CTG) — CTG will be taken from the patient's own mouth
  Arms: Tuberosity Connective Tissue Graft (CTG)

SUMMARY:
Mid-facial recession following immediate implant placement (IIP) in the place of a tooth poses a significant challenge for clinicians to treat. Emerging evidence shows that connective tissue graft (CTG) augmentation may mitigate the remodeling of the buccal bone crest (i.e., bone within the gum that supports the tooth), and lessen the soft tissue recession. A recent systemic review suggested a supplemental CTG grafting to IIP as a standard of care, especially for cases that have a high esthetic risk, specifically with a thin gingival biotype (i.e., thin gum tissue) and a thin buccal bone plate. The alternative option to augment the facial contour is the xenogeneic volume-stable collagen matrix (VCMX), which favors avoiding morbidity but hasn't been thoroughly investigated on IIP. Despite that IIP has attracted considerable scientific interest, the dynamic changes of the bone crest and soft tissue, especially during the early healing stage (<3 months following IIP), are little known. Recently, an ultrasonography protocol has been validated for its diagnostic value in dental implant research. High-frequency B-mode imaging and color flow and power Doppler are implemented to display the spatial relation of anatomic landmarks of peri-implant tissues and to visualize the flow velocity and blood volume, respectively. It provides a valuable real-time diagnostic tool to evaluate hard and soft tissue remodeling and tissue perfusion changes during the early healing stage around IIP, comparing CTG and VCMX grafting. Hence, the purpose of this three-arm RCT is to compare the clinical efficacy and longitudinal remodeling of hard and soft tissue around IIP among CTG, VCMX, and control (without soft tissue augmentation) group. This will be the first evidence of the longitudinal tissue changes around immediate implant, and the first RCT comparing the clinical efficacy and esthetic outcome of xenogenic soft tissue substitute (i.e., from the non-living bone of another species) to the gold standard approach (CTG) on the immediate implants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-95
* Has a single hopeless tooth in the maxillary esthetic zone (i.e., first premolar to first premolar, tooth #5-tooth #13)
* Adequate oral hygiene (i.e., full-mouth bleeding score (FMBS) and full mouth plaque score (FMPS) of less than 25%)
* Adequate tooth space to support an immediate implant placement (i.e., adequate mesiodistal space of greater than or equal to 6 mm and interocclusal space to support a non-occluding provisionalization).
* Postextraction vertical bone defect of the buccal socket wall was less than or equal to 3mm.

Exclusion Criteria:

* patients taking long-term (more than 3 months) medications affecting bone metabolism
* generalized untreated periodontitis with greater than of 30% of sites with greater than 5mm pocket depths and bleeding upon probing with a dental probe
* medical contraindications for having a surgical procedure (i.e., ASA Status of III, patient with a severe systemic disease that is not life-threatening; ASA Status of IV, a patient with a severe systemic disease that is a constant threat to life).
* history of radiotherapy in the head and neck region
* heavy smoker (greater than 10 cigarettes per day)
* pregnancy
* gingival recession before extraction in relation to the contralateral tooth.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaoping Zhang, DDS, MS, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tuberosity Connective Tissue Graft (CTG) | Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft | No Soft Tissue Augmentation
Started | 11 | 13 | 7
Completed | 2 | 8 | 2
Not Completed | 9 | 5 | 5
Not completed — Study terminated before all 6-month visit data could be collected | 9 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tuberosity Connective Tissue Graft (CTG) | Xenogeneic Volume-Stable Collagen Matrix (VCMX) Graft | No Soft Tissue Augmentation | Total
Number analyzed (Participants) | 11 | 13 | 7 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 5 | 16
  >=65 years | 5 | 8 | 2 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 3 | 14
  Male | 8 | 5 | 4 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Had an Implant That Survived 6 Months After Immediate Implant Placement Either With or Without Soft Tissue Grafting
Description: For participants that had immediate implant placement either with or without soft tissue grafting, this outcome is determined via clinical evaluation of the percentage of participants that still had their 1 implant in place after 6 months. Note: Only 1 implant was placed per participant.
Time Frame: 6 months after immediate implant placement
Measure: Count of Participants; unit: Participants
Arm/Group | Tuberosity Connective Tissue Graft (CTG) | Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft | No Soft Tissue Augmentation
Number analyzed (Participants) | 2 | 8 | 2
Participants | 2 | 8 | 2

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Tuberosity Connective Tissue Graft (CTG) | Xenogeneic Volume-Stable Collagen Matrix (VCMX) graft | No Soft Tissue Augmentation
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/8 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT05330702/Prot_SAP_000.pdf